CLINICAL TRIAL: NCT02130908
Title: A Study on the Possible Health Effects of Lean Fish, Fatty Fish and Lean Meat Intake in Non-obese Adults
Acronym: FISK1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Bergen Medical Research Foundation (Other); Skretting ASA (Unknown); Leroy Seafood Group ASA (Industry)
Responsible Party: Principal Investigator, Oddrun Anita Gudbrandsen, Researcher, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REK2011/572
Record Dates: First submitted 2014-05-01; First posted 2014-05-06 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Metabolic Disorders; Obesity
MeSH Terms: conditions — Metabolic Diseases; Obesity | interventions — bearberry, bladderwrack, borage oil, centella, fatty acid, fish oil, ginkgo biloba, melilotus, soya lecithin drug combination

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lean fish (Experimental)
  Interventions: Other: Lean fish
- Fatty fish (Experimental)
  Interventions: Other: Fatty fish
- Lean meat (Experimental)
  Interventions: Other: Lean meat

INTERVENTIONS:
Other: Lean fish — Participants consumed 150g of lean fish, five times per week for 4 weeks
  Arms: Lean fish
Other: Fatty fish — Participants consumed 150g of fatty fish, five times per week for 4 weeks
  Arms: Fatty fish
Other: Lean meat — Participants consumed 150g of lean meat, five times per week for 4 weeks
  Arms: Lean meat

SUMMARY:
This study is a pilot study to investigate whether intake of lean or fatty fish, or lean meat would affect parameters related to health in healthy non-obese adults, and will serve as basis for future calculation of group sizes in coming studies. Participants consumed 750g/week of fillets of fish or meat for 4 weeks.

Hypothesis:

High intake of either lean or fatty fish will not affect serum concentrations of lipids and inflammatory markers as well as improve glucose tolerance during the 4 week intervention period when compared to lean meat intake.

ELIGIBILITY:
Inclusion Criteria:

* adults
* non-obese
* healthy

Exclusion Criteria:

* diabetes
* diagnosed diseases of the intestine or cardiovacular system

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2011-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Changes in metabolic parameters (lipids, glucose, inflammatory markers) measured in serum | Endpoint after 4 weeks intervention

SECONDARY OUTCOMES:
Changes in body weight | Endpoint after 4 weeks intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Haukeland University Hospital, Bergen, Norway